CLINICAL TRIAL: NCT04865692
Title: Effects of Blood Flow Restriction on Clinical Outcomes in Women With Knee Osteoarthritis
Brief Title: Effects of Low Intensity Blood Flow Restriction on Clinical Outcomes in Women With Knee Osteoarthritis
Acronym: BFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 719-II
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The interventional group received resisted knee extension 20% of 1RM with blood flow restriction along with routine physical therapy.
  Interventions: Other: BFRT; Other: Routine Physical Therapy
- Control Group (Other): The Control group received routine physical therapy alone including knee isometrics and resisted knee extension
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: BFRT — Patients of Interventional group were treated with routine physiotherapy program combined with LI-BFR consist of 10 minutes' session 3 per week for 12 weeks. In order to determine the training load 20% of 1RM, participants had performed knee extension in full range with a challenging weight. After each test, participants rated their perceived exertion level on (RPE) scale to determine the difficulty of the resistance. The derived 1RM was used to determine the 20% 1RM load used for low-load training. Blood flow restriction proximal to the working muscles achieved through using pressure cuffs. The cuff was applied to the proximal thigh. During week 1 the inflation pressure was 100mmHg. Final exercise pressure based the week of the training. Quadriceps size was measured by tape measures thigh
  Arms: Interventional group
Other: Routine Physical Therapy — knee isometrics, resisted knee extension with chalanging weight 2 sets of 10 Reps with 5 sec hold

SUMMARY:
Objective is to compare the effects of routine physical therapy with and without low intensity blood flow restriction on pain and quadriceps muscle strength in women with knee osteoarthritis.

A single blinded randomized controlled trial conducted at Department of Physiotherapy, University of Lahore Teaching Hospital, Defense Road, Lahore.

Total 60 participants were randomly assigned in to two groups, with 30 in each group The intervention group received routine physiotherapy program combined with Low Intensity Blood Flow Restriction Technique (LI-BFR. While control group were treated with only routine physiotherapy.

Dynamometer was used to assess the knee extensor strength while Knee injury and osteoarthritis outcome score was used to record any exacerbation in pain and effects of BFR on activities of daily living. Training load determined 20% of 1RM. Data analysis had done on SPSS version 23.

DETAILED DESCRIPTION:
nonparametric test Friedman test was for comparison within the groups and Mann Whitney U test was used for comparison between groups.

Randomization had done through the sealed envelope method. After allocation subjects had received their treatment protocals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients of grade II knee osteoarthritis
* Patient's age 45-65

Exclusion Criteria:

* Bilateral knee replacement
* Lower limb surgery in the last six months
* Diagnosis of inflammatory joint or muscle disease
* Chest pain during exercise or at rest; or need for supplemental oxygen
* Pregnancy
* Any systemic disease

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle strength | 12 Weeks
  dynamometer was used to assess strength
thigh muscle size | 12 weeks
  measuring tape was used to measure
Pain | 12 weeks
  pain was measured through NPRS

SECONDARY OUTCOMES:
Activities of daily living | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: zoya Mujahid, DPT, Study Chair — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No